CLINICAL TRIAL: NCT06099379
Title: Modulation of ∆9-tetrahydrocannabinol Acute Psychoactive Effects by Ranging Doses of Cannabidiol in Healthy, Occasional Cannabis Users: a Controlled, Triple Blind, Randomized, Cross-over Study
Brief Title: Modulation of THC Effects by CBD: a Dose-ranging Study
Acronym: SPECTRE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 2024-11772
Record Dates: First submitted 2023-09-29; First posted 2023-10-25 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Cannabis; THC
MeSH Terms: conditions — Marijuana Abuse | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: In this crossover design, participants will be administered all phytocannabinoid doses contained in the four CBD:THC products and the control product (THC only) during participation in the study. Participant will be randomly assigned to one of the predetermined sequences with a CBD:THC product or control product at 5 dosages (CBD:THC of 0:20 mg, 20:20 mg, 40:20 mg, 80:20 mg and 120:20 mg). Participants will be randomized based on a balanced 5 by 5 Latin square.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- CBD:THC Group 1 (Experimental): Group will receive four doses of CBD:THC ratio (20:20 mg, 40:20 mg, 80:20 mg and 120:20 mg) and a control product CBD:THC ratio (0:20 mg).
  Group will attend a total of five study visits (one for each study product) with at least 1 week between each visit.
  The order in which the study products will be administered depend on the randomization sequence.
  Interventions: Drug: ∆9-tetrahydrocannabinol
- CBD:THC Group 2 (Experimental): Group will receive four doses of CBD:THC ratio (20:20 mg, 40:20 mg, 80:20 mg and 120:20 mg) and a control product CBD:THC ratio (0:20 mg).
  Group will attend a total of five study visits (one for each study product) with at least 1 week between each visit.
  The order in which the study products will be administered depend on the randomization sequence.
  Interventions: Drug: ∆9-tetrahydrocannabinol
- CBD:THC Group 3 (Experimental): Group will receive four doses of CBD:THC ratio (20:20 mg, 40:20 mg, 80:20 mg and 120:20 mg) and a control product CBD:THC ratio (0:20 mg).
  Group will attend a total of five study visits (one for each study product) with at least 1 week between each visit.
  The order in which the study products will be administered depend on the randomization sequence.
  Interventions: Drug: ∆9-tetrahydrocannabinol
- CBD:THC Group 4 (Experimental): Group will receive four doses of CBD:THC ratio (20:20 mg, 40:20 mg, 80:20 mg and 120:20 mg) and a control product CBD:THC ratio (0:20 mg).
  Group will attend a total of five study visits (one for each study product) with at least 1 week between each visit.
  The order in which the study products will be administered depend on the randomization sequence.
  Interventions: Drug: ∆9-tetrahydrocannabinol
- CBD:THC Group 5 (Experimental): Group will receive four doses of CBD:THC ratio (20:20 mg, 40:20 mg, 80:20 mg and 120:20 mg) and a control product CBD:THC ratio (0:20 mg).
  Group will attend a total of five study visits (one for each study product) with at least 1 week between each visit.
  The order in which the study products will be administered depend on the randomization sequence.
  Interventions: Drug: ∆9-tetrahydrocannabinol

INTERVENTIONS:
Drug: ∆9-tetrahydrocannabinol — Phytocannabinoids from plant inflorescences (CBD and THC dominant) - inhaled
  Other Names: Cannabidiol

SUMMARY:
The purposes of this study are 1) to determine if CBD modulates THC-induced acute psychoactive effects at different CBD:THC ratios, compared with the control product (0:20, 20:20, 40:20, 80:20, 120:20) and 2) to determine if different doses of CBD modulate other THC induced behavioral effects, compared with the control product and 3)To explore qualitatively whether CBD modulates THC effects by mechanisms that are not detected with standard clinical research tools.

DETAILED DESCRIPTION:
Despite more than 40 years of research on the active compounds present in the cannabis plant, the influence of CBD consumption on the metabolism, pharmacology, and behavioral effects of THC remains fragmentary and scarcely documented in vivo in humans. Cannabis users are currently encouraged to choose products containing CBD, but evidence is lacking regarding its potential benefits when consumed jointly with THC across different ratios. Given the recent cannabis legalization in Canada and the widespread use of inhalation as the preferred mode of administration for non-therapeutic cannabis, closing this knowledge gap will help ensure public safety and allow regulatory bodies and public health authorities to elaborate more refined cannabis use guidelines and harm reduction strategies. It will also empower people who use cannabis to make more informed purchasing decisions and will drive the incubation of future research endeavors in the fields of medical and social sciences. The aim of this study is to improve our understanding of the (acute) behavioral and pharmacological effects of different doses of CBD administered concomitantly with THC via inhalation in individuals who engage in occasional cannabis use, taking into consideration multiple factors that can modulate such effects. This study will put to the test conceptions surrounding the interaction between specific cannabinoids by evaluating the role of CBD on the modulation of THC's effects pertaining to cognition, behavior, subjective experience, and physiological parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Between 21 and 49 years of age, inclusively;
2. Have used cannabis at least once in their lifetime and have used cannabis three days or less in the 30 days prior to enrollment;
3. Be able to provide a signed informed consent;
4. Willing to comply with study procedures and requirements as per protocol;
5. Have a forced expiratory volume in first second (FEV) less than or equal to 90 %;
6. Able to communicate and understand English or French language;
7. For female participants:

   a. No childbearing potential, defined as: i. postmenopausal (12 months of spontaneous amenorrhea and ≥ 45 years of age); or ii. Documented surgically sterilized (i.e., tubal ligation, hysterectomy, or bilateral oophorectomy); or b. For female of childbearing potential: i. Must have negative pregnancy test result at screening and at subsequent visits.

ii. AND have no pregnancy plan while on the study iii. AND must agree to use a medically accepted method of birth control throughout the study.

Exclusion criteria

Participants will be excluded if any of the following criteria are met:

1. Any disabling medical condition, as assessed by medical history, physical exam, vital signs and/or laboratory assessments that, in the opinion of the study physician, precludes safe participation in the study or the ability to provide fully informed consent;
2. Severe psychiatric condition (history of schizophrenia, schizoaffective disorder or bipolar disorder; current acute psychosis, mania or current suicidality based on the Mini International Neuropsychiatric Interview);
3. Any other disabling, unstable or acute mental condition that, in the opinion of the study physician, precludes safe participation in the study or ability to provide fully informed consent;
4. Known chronic liver disease or aspartate transaminase/alanine transaminase (AST/ALT) two times higher than upper limit of normal values at screening visit;
5. Blood pressure higher than 130/80 mmHg;
6. Kidney disorders;
7. Bleeding disorders;
8. Current moderate or severe DSM-5 substance use disorder (except nicotine) according to SCID-V;
9. Currently pregnant, breastfeeding or planning to become pregnant either at screening or while enrolled in the study;
10. Pending legal action or other reason that, in the opinion of the study physician, might prevent study completion;
11. Use of medication within 7 days of experimental sessions; which, in the opinion of the Investigator, may interact with cannabis.
12. Participation in clinical studies or undergoing other investigational procedure involving cannabis or cannabinoids administration within 30 days prior to randomization.
13. Resting heart rate over 100 beats per minute.
14. Current body mass index (BMI) over 29.9 kg/m2.
15. Any clinically significant electrocardiogram abnormalities at screening visit.

Ages: 21 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective and subjective measures of cannabinoids effect | Prior to the Product administration ,10 minutes and 80 minutes after inhalation
  Based on the scores obtained on the observer items (objective) and the participant-rated items (subjective) from the Clinician Administered Dissociative State Scale (CADSS). The CADSS is a 28-item validated instrument, includes 5 observer items and 23 participant self-report items rated on a 5-point scale, ranging from 0 (not at all) to 4 (extremely) on eight items. The score will reflect the extent to which participants were observed to be under the effect of cannabinoids, i.e., in adissociative state.

SECONDARY OUTCOMES:
Positive and Negative Affect | Prior to the Product administration , 10 minutes and 80 minutes post inhalation
  Will be measured by the Positive and Negative Affect Schedule (PANAS). The PANAS is a 20-item validated questionnaire, used in both non-clinical and clinical populations.
Neural oscillations | Prior to the Product administration, 80 minutes post inhalation and at the end of the study visit, approximatively 140 minutes after inhalation
  Auditory oscillations, using an electroencephalogram (EEG), will be probe in response to 40-Hz FM and ascending/descending AM stimuli, using a 16-channel system with 250-Hz sampling rate and 24-bit resolution (model g.Nautilus PRO 16 g.SAHARA, g.tec, Schiedlberg, Austria).
Anxiety Symptoms | Prior to the Product administration, 10 minutes and 80 minutes after inhalation
  Symptoms of anxiety will be assessed using the States-Trait-Anxiety-Inventory (STAI). It consists of two 20-item self-report scales (trait and state anxiety) that measure the severity of anxiety in adults. Both subscales are composed of 20 statements rated on a 4-point Likert scale ranging from 1 ("not at all" and "almost never" for the state and trait subscales, respectively) to 4 ("very much" and "almost always" for the state and trait subscales, respectively).
Subjective Drug Effects | 10 minutes and 80 minutes after inhalation
  Drug Effect Questionnaire (twenty-three-item) will be use to assess participant's physical signs, symptoms associated with cannabis inhalation and desire to use the product. The Drug Effects Questionnaire uses visual analogue scale, ranging from 0 (not at all) to 100 (extremely).
Experience with Study Products | 140 minutes after inhalation
  Subjective effects of cannabis will be assessed using the Cannabis Experience Questionnaire (CEQ), The CEQ measures participants' subjective experiences with cannabis consumption and consists of two subscales: pleasurable experiences (18 items), psychosis-like experiences (25 items), and after-effect experiences measuring the consequences of cannabis after use (12 items). Each item of each subscale is rated on a 5-point Likert scale, ranging from 1 (not at all) to 5 (extremely).
Social Exposition Challenge | 70 minutes after inhalation
  This will help determine if different doses of CBD can modulate the feeling of paranoia and/or anxiety triggered by social interactions, in comparison to the control product. The research staff will give to the participant five dollars in cash. The participant will then be escorted out of the research center by a member of the research staff for a 10-minute walk to the hospital pharmacy with the instruction of purchasing an item of their choosing with the money. Once the task is completed, the participant will be escorted back to the research center. The research staff will walk approximately two meters behind the participant during the whole procedure and will be instructed not to engage in any conversation, unless the participant needs assistance or feels abnormally anxious.
Change on cognition | Prior to the Product administration (only at Visite 1) and 10 minutes after inhalation at each visit
  The Cambridge Neuropsychological Test Automated Battery tests will be used for the rapid assessment of multiple cognitive components.
Success of Blinding Questionnaire | 10 minutes and 140 minutes after inhalation
  To assess the success of the blind iwith the Blinding Success Questionnaire (BSQ). The specific aims of testing the blind are to a) determine which research product participants think they received and b) examine the associations between the research product participants think they received and their expectations, subjective cannabis perceptions, treatment outcomes, and side effects.
Inhalation Adherence | During inhalation procedure
  When the participant inhales the investigational product, research staff will fill a questionnaire assessing participant compliance.
Change in Safety | Baseline,10 minutes, 80 minutes and 140 minutes after inhalation
  Adverse events will be collected prior to administration of the study product (T0) and following administration of the study product (T1, T2 and T3).
Visit Intoxication Assessment | Through study visit completion, approximatively 140 minutes after product inhalation
  Signs of intoxication will be assess using the modified Standardized Field Sobriety Test.

OTHER OUTCOMES:
Change in plasma concentrations of CBD | Prior to the Product administration and 5,15, 80, 110, and 140 minutes after administration
  Plasma levels of CBD will be determined by high performance liquid chromatography-tandem mass spectrometry.
Change in plasma concentrations of THC | Prior to the Product administration and 5,15, 80, 110, and 140 minutes after administration
  Plasma levels of THC will be determined by high performance liquid chromatography-tandem mass spectrometry.
Change in plasma concentrations of Anandamide (AEA) | Prior to the Product administration and 5,15, 80, 110, and 140 minutes after administration
  Plasma levels of CBD and THC will be determined by high performance liquid chromatography-tandem mass spectrometry.
Change in plasma concentrations of 2-Arachidonoylglycerol (2-AG) | Prior to the Product administration and 5,15, 80, 110, and 140 minutes after administration
  Plasma levels of CBD and THC will be determined by high performance liquid chromatography-tandem mass spectrometry.
Genetic markers | Baseline, Prior to the Product administration (only at visite 1)
  To explore potential genetic factors that could explain at least in part some of the participants' responses to the study outcomes and that have been associated with specific candidate genes (e.g., COMT, AKT1, DRD2, FAAH and cytochrome P450 genes). Using buccal swabs from EndoDNA test kits. These DNA tests will be used to map known genetic variants associated with the endocannabinoidome and related physiological systems to identify specific genotypes that correlate with neurocognitive and behavioral effects measured for each study product for an example application of the method).

CONTACTS AND LOCATIONS:
Overall Officials: Didier Jutras-Aswad, MD, MS, Principal Investigator — CRCHUM
Locations (1):
- Centre de recherche du Centre Hospitalier Universitaire de Montréal, Montreal, Quebec, Canada